CLINICAL TRIAL: NCT01512342
Title: Pacing Activity Self-management for Patients With Chronic Fatigue Syndrome: Randomized Controlled Clinical Trial
Brief Title: Pacing Activity Self-management for Patients With Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Artesis University College, Antwerp (Other); Universiteit Antwerpen (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Jo Nijs, Associate professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PacingCFS; Artesis University College (Other: Artesis University College Antwerp)
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Fatigue Syndrome
Keywords: pacing; activity management; relaxation; physiotherapy; occupational therapy; autonomic nervous system
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pacing (Experimental): The pacing self-management program focussed on teaching the patient to estimate their current physical capabilities prior to commencing an activity. In order to appropriately pace activities (daily activities and exercise bouts), CFS patients were learned to estimate their current physical capabilities prior to commencing an activity, keeping in mind the regular fluctuating nature of their symptoms. The activity duration used within the program was less than that reported by the patient so to account for typical overestimations made by the patient. Each activity block was interspersed with breaks, with the length of this break equating to the duration of the activity.
  Interventions: Behavioral: Pacing
- relaxation therapy (Active Comparator): Relaxation therapy comprised of education about the role of stress in CFS biology, and the opportunities stress management provides to handle this issue. Patients were then taught how to apply stress management techniques like Jacobson relaxation skills, Schultz relaxation skills, visualization, etc.
  Interventions: Behavioral: relaxation therapy

INTERVENTIONS:
Behavioral: Pacing — 3 one-on-one sessions weekly for 3 consecutive weeks
  Other Names: activity self-management; activity management; adaptive pacing
  Arms: Pacing
Behavioral: relaxation therapy — 3 one-on-one sessions weekly for 3 consecutive weeks
  Other Names: stress managament; Jacobson relaxation; visualisation; Schultz relaxation
  Arms: relaxation therapy

SUMMARY:
Given the lack of evidence in support of pacing self-management for patients with chronic fatigue syndrome (CFS), it is examined whether physical behavior and health status of patients with CFS improve in response to a pacing self-management program. The effects of pacing will be compared with those observed when applying relaxation therapy to patients with CFS.

DETAILED DESCRIPTION:
Given the lack of evidence in support of pacing self-management for patients with chronic fatigue syndrome (CFS), it is examined whether physical behavior and health status of patients with CFS improve in response to a pacing self-management program. The effects of pacing will be compared with those observed when applying relaxation therapy to patients with CFS.

According to the power calculation, 36 patients fulfilling the 1994 Centre for Disease Control and Prevention criteria for the diagnosis of chronic fatigue syndrome (CFS) will be randomized to either 3 weeks of pacing activity self-management or relaxation therapy. Both treatment groups will receive 3 weekly sessions spread over 3 consecutive weeks. All treatments will be delivered by occupational therapists or physiotherapists. One treatment session lasts for about 45 minutes each.

Outcome measures include the Canadian Occupational Performance Measure (COPM), Medical Outcomes Short Form 37 Health Status Survey (SF-36), Checklist Individual Strength (CIS), CFS Symptom List and autonomic activity at rest and following 3 activities of daily living (writing a standardized test on a laptop computer, ironing, and climbing 26 flights of stairs). For measuring autonomic activity, the Nexus 10 device (Mind Media, the Netherlands) will be used. Skin conductance, body temperature, heart rate, blood volume pressure and heart rate variability will be measured continuously in real time during a 2 minutes period, with the patient sitting on a chair (back supported and hands resting on legs). Electrodes will be placed on the left hand in all patients.

ELIGIBILITY:
Inclusion Criteria:

* adult
* age range between 18 and 65 years of age
* female gender
* willing to sign informed consent form
* fulfilling the 1994 Centre for Disease Control and Prevention criteria for the diagnosis of chronic fatigue syndrome

Exclusion Criteria:

- Not fulfilling each of the inclusion criteria listed above.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
the change in score on the Canadian Occupational Performance Measure (COPM) | measured at baseline (week 1) and post-treatment (week 5)
  well-validated, reliable and frequently used outcome measure semi-structered interview

SECONDARY OUTCOMES:
the change in subscale scores on the Medical Outcomes Short Form 37 Health Status Survey (SF-36) | measured at baseline (week 1) and post-treatment (week 5)
  The SF-36 assesses functional status and well-being or quality of life. The SF-36 has been documented to have reliability and validity in a wide variety of patient populations and it is the most frequently used measure in CFS research.
the change in Ckecklist Individual Strength (CIS) | measured at baseline (week 1) and post-treatment (week 5)
  The CIS aims at assessing the subjective fatigue experience, concentration difficulties, motivation and physical activity. Higher scores on the CIS correspond to severe fatigue, many concentration difficulties, problems with motivation and a low level of physical activity. Its psychometric properties are well established.
the change in CFS Symptom List | measured at baseline (week 1) and post-treatment (week 5)
  The CFS Symptom List is a self-reported measure for assessing symptom severity in CFS patients. In order to assess the severity of the symptoms included in the CFS Symptom List, visual analogue scales (100 mm) are used. Psychometric work supporting the use of the CFS Symptom List has been published.
the change in autonomic activity at rest and following 3 activities of daily living | measured at baseline (week 1) and post-treatment (week 5)
  The 3 activities of daily living entail writing a standardized test on a laptop computer, ironing, and climbing 26 flights of stairs. For measuring autonomic activity, the Nexus 10 device (Mind Media, the Netherlands) will be used. Skin conductance, body temperature, heart rate, blood volume pressure and heart rate variability will be measured continuously in real time during a 2 minutes period, with the patient sitting on a chair (back supported and hands resting on legs). Electrodes will be placed on the left hand in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Kos, PhD, Study Director — Artesis University College Antwerp, Belgium
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

REFERENCES:
- [Background] Nijs J, van Eupen I, Vandecauter J, Augustinus E, Bleyen G, Moorkens G, Meeus M. Can pacing self-management alter physical behavior and symptom severity in chronic fatigue syndrome? A case series. J Rehabil Res Dev. 2009;46(7):985-96. doi: 10.1682/jrrd.2009.01.0007. PMID 20104421
- [Background] Nijs J, Paul L, Wallman K. Chronic fatigue syndrome: an approach combining self-management with graded exercise to avoid exacerbations. J Rehabil Med. 2008 Apr;40(4):241-7. doi: 10.2340/16501977-0185. PMID 18382818
- [Background] Meeus M, van Eupen I, van Baarle E, De Boeck V, Luyckx A, Kos D, Nijs J. Symptom fluctuations and daily physical activity in patients with chronic fatigue syndrome: a case-control study. Arch Phys Med Rehabil. 2011 Nov;92(11):1820-6. doi: 10.1016/j.apmr.2011.06.023. PMID 22032215
- [Derived] Larun L, Brurberg KG, Odgaard-Jensen J, Price JR. Exercise therapy for chronic fatigue syndrome. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD003200. doi: 10.1002/14651858.CD003200.pub9. PMID 39697147
- See also: International Pain in Motion research group — http://www.paininmotion.be